CLINICAL TRIAL: NCT06723119
Title: The Effects of Resveratrol Supplementation on Functional and Systemic Markers of Muscle Damage and Cardiovascular Function in Response to a Damaging Isoinertial Squat Protocol
Brief Title: Effect of Resveratrol Supplementation on Exercise Performance and Recovery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Central Florida (Other)
Collaborators: Gencor Pacific Group (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00006703
Record Dates: First submitted 2024-11-20; First posted 2024-12-09 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-11

CONDITIONS: Effect of Resveratrol on Performance and Recovery
MeSH Terms: interventions — Resveratrol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Resveratrol Supplementation (Active Comparator): Once daily (immediately upon waking) supplementation with 500mg (2 capsules) VeriSperse® resveratrol (VRES) for 17 days
  Interventions: Other: Resveratrol (VRES) 500 mg oral once daily.
- Placebo (Placebo Comparator): Once daily (immediately upon waking) supplementation with 500mg (2 capsules) Placebo (maltodextrin) for 17 days
  Interventions: Other: Placebo 500 mg oral once daily.

INTERVENTIONS:
Other: Resveratrol (VRES) 500 mg oral once daily. — Resveratrol supplement will be provided in capsule form within a distinctly labeled bottle. Participants will be instructed to consume 2 capsules (500mg) of their assigned supplement with at least 8oz of water immediately upon waking for 17 days.
  Arms: Resveratrol Supplementation
Other: Placebo 500 mg oral once daily. — Placebo will be supplement will be provided in capsule form within a distinctly labeled bottle. Participants will be instructed to consume 2 capsules (500mg) of their assigned supplement with at least 8oz of water immediately upon waking for 17 days.
  Arms: Placebo

SUMMARY:
To examine the effects of once daily supplementation with 500mg VeriSperse® resveratrol (VRES) for 17 days on muscle function, delayed onset muscle soreness, systemic concentrations of muscular damage markers and markers of oxidative stress in resistance trained young adult males following a damaging isoinertial squat protocol (ISP).

DETAILED DESCRIPTION:
This study will utilize a randomized counter balanced cross-over repeated measures design. Participants will complete a total of 13 visits to the Exercise Physiology Intervention and Collaboration (EPIC) lab.

6.2 Procedures of each individual visit: Visit 1 (V1): will consist of informed consent and eligibility screening. Individuals who have provided written informed consent to participate will be screened using the Physical Activity Readiness Questionnaire (PAR-Q+), Medical History Questionnaire (MHQ), and a Caffeine Consumption Questionnaire (CCQ) to determine eligibility to participate in the study. Eligible participants will also be examined by a certified phlebotomist to determine the likelihood of successful venipuncture. Eligible participants will subsequently be randomized in a counter balanced fashion into two treatment groups (n=10/group) corresponding to either Verisperse® Resveratrol (VRES) or Placebo (PLA) using an online randomization tool. Participants will also select their snack choice from a list of pre-approved options. Following this, participants will be scheduled for visit 2 (V2), which will occur at least 24 hours following V1.

Visit 2 (V2): Participants will arrive for V2 in a fasted state (≥8 hours) having abstained from alcohol for at least 12 hours prior. Upon arrival, participants will complete a hydration assessment by urinating into a provided sample cup no more than 4oz. Participants will then provide a venous blood sample to determine baseline systemic concentrations of creatine kinase and C-reactive protein. Next, participants will complete anthropometric assessments of height, weight, and body composition via bioelectrical impendence analysis (BIA). Participants will be asked to remove shoes and all jewelry for BIA. There are no risks or discomfort associated with the bioelectrical impendence analysis. Next, participants will be rested in a quiet, dimly lit laboratory in a semi-recumbent position for 15 minutes before completing the flow-mediated dilation (FMD) assessment. Participants will then be provided with their standardized snack of choice (energy bar) before undergoing familiarization with the active range of motion (AROM), pain pressure threshold (PPT), muscle soreness (MS) perceived recovery scale (PRS), maximal voluntary isometric contraction (MVIC), and vertical jump (VJ) assessments and the isoinertial squat protocol (ISP) (3 sets of 6 repetitions at a resistance of .067kg/mm2). Following the ISP, participants will be familiarized with the online MyFitnessPal application.

Visits 3-5 (V3-V5): Upon arrival for V3-V5, participants will undergo a standardized warm-up identical to V2 before completing additional familiarization with the ISP. All procedures for V3-V5 will be identical. V2-V5 will be separated by at least 24-hours but no more than 72 hours.

Visit 6 (V6): Upon arrival to the lab participants will fill out a sleep quality questionnaire (SQQ), provide a urine sample to assess hydration status, and provide a pre-exercise venous blood sample to establish baseline measures of creatine kinase (CK) and C-reactive protein (CRP). Next, participants will complete PRE ultrasound assessments of muscle thickness (MT) and echo intensity (EI) followed by the FMD assessment. Participants will then be provided with the standardized snack (energy bar) of their choice and complete a standardized warmup identical to V2, before completing PRE assessments of AROM, PPT, MS, PRS, MVIC, and VJ. Participants will then be fitted with a heart rate monitor and complete the ISP followed by a 3-minute cycle-based cool down period, a venous blood sample, and follow-up assessments of MT, EI, AROM, PPT, MS, PRS, MVIC, and VJ immediately post-exercise (IP). MVIC and VJ will be separated by 5 minutes to allow for adequate recovery.

Visits 7-9 (V7-V9): V7-V9 will be identical in nature and will occur 24, 48, and 72 hours following V6, respectively. Upon arrival to the lab for each experimental trial (V7-V9) participants will fill out a sleep quality questionnaire (SQQ), provide a urine sample to assess hydration status, and provide a pre-exercise venous blood sample to establish baseline measures of creatine kinase (CK) and C-reactive protein (CRP). Next, participants will complete ultrasound assessments of muscle thickness (MT) and echo intensity (EI) followed by the FMD assessment. Participants will then complete a standardized warmup identical to V2, before completing assessments of AROM, PPT, MS, PRS, MVIC, and VJ. MVIC and VJ will be separated by 5 minutes to allow for adequate recovery.

Visit 10 (V10): V10 will occur 32 days after V9 and be conducted in an identical fashion to V6.

Visits 11-13 (V11-V13): V11-V13 will occur 24, 48, and 72 hours following V10, respectively. V11-V13 will be conducted in an identical fashion to V7-V9)

Consent and Screening Prior to beginning the study, individuals interested in participating in the study will be asked to report to the EPIC lab to review and sign an informed consent document. Participants who provide consent to participate will then be screened for eligibility via the PAR-Q+, MHQ, and CCQ. Participants will also be asked to fill out a contact form that will record their preferred email and cell phone number.

Hydration Status Assessment Upon arriving to the lab, participants will be given a sample cup to take to the restroom and provide a urine sample, so that hydration may be assessed. After providing a urine sample, a member of the research team will measure urine specific gravity (USG) using a refractometer to ensure participants are euhydrated (1.002-1.025). If dehydrated (>1.025), they will be asked to consume 16 oz of water and be retested after waiting 15 minutes post ingestion. If hyperhydrated (<1.002) their visits will be rescheduled. Hydration status will be checked immediately upon arrival to the laboratory for V2 and each experimental trial (V6-V13). Urine samples will be disposed of according to UCF policy.

Venous Blood Sample Collection Blood samples at V2, PRE-, IP, 24H, 48H, and 72H will be obtained using a 21-gauge, 1¼ inch vacutainer blood collection needle or 23-gauge butterfly needle taken from a superficial forearm vein. A maximum of 2 unsuccessful attempts to insert a needle in one of the participant's arms will be made and, with their permission, a third and final attempt will be made in the opposite arm. Three unsuccessful venipuncture attempts will result in termination of the blood draw. Issues with blood collection devices that prevent the drawing of blood are not grounds for removal from the study and will not affect participants continuation with the remainder of the study. All blood draws will be conducted under aseptic conditions. To minimize the risks, the skin area where the needle is inserted will be cleaned and prepared with a disinfectant alcohol wipe before the needle is inserted. Following the blood draw, the puncture site will be covered with a bandage.

A total of 8mL (slightly less than 2 tsp) of blood will be collected at each time point (V2 & V6-V13) in one 4mL BD Vacutainer™ Serum separation tube (SST) and one 4mL K2EDTA plasma tube (EDTA).

Blood samples collected in the 4mL SST tube will be used to determine serum concentrations of C-reactive protein (CRP) and creatine kinase (CK). Serum tubes will be inverted ten times and allowed to clot at room temperature for 30-minutes prior to centrifugation for 10-minutes at 4000rpm. After centrifugation, serum will be aliquoted and frozen at -80°C within one hour of collection.

Blood samples collected in EDTA tube will be gently inverted ten times and left at room temperature for same day analysis. EDTA whole blood samples will be analyzed directly in-house using an automated hematology analyzer (Sysmex XN-450 Automated Hematology Analyzer) located in the Cellular Exercise Physiology Laboratory (CEPL) in BIO 224, Building 20 (Biological Sciences). Sample analytes will include hematocrit, hemoglobin, mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), and total (white blood cell and red blood cell) and differential (lymphocyte, monocyte, and granulocyte, platelet) cell counts.

Standardized Warm-up Prior to all performance assessments, participants will be required to complete a dynamic warm-up. Participants will begin by pedaling on a cycle ergometer for 5-minutes at a self-selected pace at a set resistance of 75 watts. Participants will then complete ten body-weight squats, ten body-weight walking lunges, ten dynamic straight leg kicks, and ten dynamic walking quadricep stretches.

Sleep Quality Questionnaire Participants will be asked to fill out a brief 7 question sleep questionnaire consisting of questions pertaining to their sleep and sleep quality within the last 24 hours. Participants will complete the SQQ immediately upon arriving for each experimental trial (V6-V13) Diet and Dietary Log Participants will be asked to maintain two separate 5-day dietary logs using the "MyFitnessPal" application on their own cellular or computer device. Participants will be asked to begin each 5-day log 24 hours before ET1 and ET2 and to maintain the log by tracking all food and beverage consumption to the best of their ability for the 5 days until the completion of the 72H follow up visits (visits 9 & 13, respectively). Additionally, participants will be asked to keep their food and beverage consumption during the two 5-day periods as consistent as possible and to match macronutrient (fats, carbohydrates, and proteins) consumption between the two periods to the best of their ability. Participants refusing to voluntarily report food and beverage consumption will be withdrawn from the study.

Assessments Anthropometric Assessments: During V2, participants will complete anthropometric assessments of height, weight, and body composition. Height and weight will be assessed using a stadiometer and scale (Health-o-meter Professional Patient Weighing Scale, Model 500 KL, Pelstar, Alsip, IL, USA). Body composition will be assessed using bioelectrical impedance analysis (BIA; InBody 770, Biospace Co, Ltd. Seoul, Korea) or bioelectrical impedance spectroscopy analyzer (Sozo; Carlsbad, CA, USA). Participants will be asked to void their bladder, and remove shoes, socks, and all jewelry for this assessment. They will also be asked to be eight hours fasted and well-hydrated as determined by USG analysis. There are no risks or discomforts associated with the BIA analysis.

Flow Mediated Dilation (FMD) Standardization of FMD procedures and protocol will be conducted following established guidelines (40). Prior to testing, subjects will be rested in a quiet, dimly lit laboratory in a semi-recumbent position for 15 minutes. Automated brachial artery sphygmomanometry (IntelliSense® Professional Monitor, OMRON Healthcare Inc., Lake Forest, IL) will be used to measure resting systolic blood pressure (SBP), diastolic blood pressure (DBP) and heart rate (HR) on the left arm. Mean arterial pressure (MAP) will be calculated to determine peripheral vascular resistance using the following equation: {MAP=[0.33×(SBP-DBP)]+DBP}. Brachial artery diameter and blood velocity will be measured by duplex, high-resolution Doppler ultrasound (GE Logiq P9, GE Healthcare, Chicago, IL) using a (5)-MHz linear array transducer. An arm tourniquet cuff with rapid inflation system (Hokanson E20; D.E. Hokanson Inc., Bellevue, WA) will be placed around the right forearm, immediately distal to the antecubital fossa for assessment of reactive hyperemia and brachial artery FMD. Stable imaging of the brachial artery will be accomplished using foam positioning aids and transducer stabilizing clamp.

Brachial artery FMD will be continuously measured and recorded using a 10-minute protocol. Baseline diameter and blood velocity will be recorded for two minutes. The tourniquet cuff will then be inflated to approximately 240 mmHg to occlude the brachial artery for five minutes. Following cuff deflation, recording will continue for three minutes to assess changes in diameter and blood velocity. All ultrasound settings will be kept consistent, and measurement will be completed by the same technician (Mr. Dufner). Scans will be recorded directly from the ultrasound system using commercial video capturing software (Snagit, TechSmith Corp., Michigan, USA) and saved to an online file drive. Offline analyses will be performed using edge-detection and wall-tracking software (FMD Studio, Cardiovascular Suite, Quipu, Pisa). Following data processing, all macro- and micro-vascular function parameters will be calculated using a custom visual basic macro in Microsoft Excel (3). FMD will be assessed during V2 and at PRE, 24H, 48H, and 72H during each experimental trial.

Ultrasound Measurement (MT and EI) Rectus femoris (RF), vastus medialis (VM) and vastus lateralis (VL) MT and EI assessments will be taken on the right leg using B-mode ultrasound (GE Logiq, General Electric Medical Systems, Milwaukee, WI, USA) and a linear array probe (L4-12t, 4.2-13.0 MHz, 38.4-mm field of view, GE Healthcare, Milwaukee, WI, USA). All ultrasound measurements will be performed at 12 MHz, gain of 50 dB, depth of 5cm, and Dynamic range of 72. A water-soluble transmission gel will be applied to the skin to enhance acoustic coupling. Three images of each muscle will be captured in the sagittal plane. RF images will be captured at half the distance between the superior border of the patella and the center of the inguinal fold. VM images will be captured between the center of the inguinal fold and 3 inches proximal to the medial epicondyle of the femur. VL images will be captured at half the distance between the greater trochanter and the superior border of the patella. Ultrasound images will be analyzed using ImageJ software (Version 1.53v., National Institutes of Health, Bethesda, MD, USA), according to the procedures described by Girts. Et al. (41). MT and EI will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Active Range of Motion (AROM) AROM will be assessed following the standardized warm-up while participants are in a prone position on a padded testing table with their legs fully supported. A handheld goniometer will be used to assess AROM of the right knee. The goniometer will be anchored at the lateral epicondyle of the femur with the stationary arm in line with the greater trochanter of the femur and the movement arm aligned with the lateral malleolus of the ankle. Participants will be instructed to move the knee from maximal full extension throughout the range of motion to maximum full flexion holding each end point for two seconds. The average of two consecutive measurements will be used to determine AROM. AROM will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Pain Pressure Threshold PPT will be assessed immediately following the AROM assessment while the participants sat on the end of padded table with their upper legs supported and their lower legs hanging freely. Using a handheld 15kg dolorimeter with a 1 cm rubber tip, pressure will be applied to the RF, VM, and VL at locations identical to that of the ultrasound assessments increasing at a rate of 1 kg/s until participants first report feeling pain, at which point the algometer will be removed from the skin. PPT will be assessed once at each sight before a second measure of PPT at each location is acquired. The algometer value at the onset of pain will be recorded and the average of two measures with will be used to denote PPT. PPT will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Perceived Recovery Scale (PRS) PRS will be assessed as a total feeling of recovery in the lower extremities (waist down) and be performed while the participant is standing at a knee angle of 140 degrees immediately prior to MS testing. Participants will be asked to rank their level of recovery on a 100mm VAS ranging from 0 to 100, with 0 being not at all recovered and 100 being very well recovered. PRS will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Muscle Soreness (MS) MS will be assessed as a total feeling of soreness in the lower extremities (waist down) and be performed while the participant is standing at a knee angle of 140 degrees immediately prior to MVIC testing. Participants will be asked to rank their level of MS of their entire lower extremities on a 100mm VAS ranging from 0 to 100, with 0 being no pain at all and 100 being the most pain imaginable. MS will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Maximal Voluntary Isometric Contraction (MVIC) and Rate of Force development (RFD) MVIC assessments will be completed inside a specialized isometric squat rack and platform with an immovable bar. Bar height for each participant will be set at a height that elicits a participant knee angle of 140 degrees. Bar height will be established during V2 and standardized for all subsequent MVIC assessments. Each MVIC assessment will consist of 3 x 5s maximal isometric contractions. For each contraction, participants will be instructed to drive upwards maximally against the bar by extending their knees and hips for 5s in a manner identical to the movement pattern of a typical high bar back squat. Each contraction will be initiated following a verbal prompt from the researcher and consistent verbal encouragement will be provided for the entire 5s of each contraction. One minute of rest will be provided between each contraction to allow for recovery. The contraction containing the highest peak force will be denoted as the participant's MVIC from which rate of force development (RFD) will be recorded at 0-250ms, dictated by the onset of muscular contraction. MVIC and RFD will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Vertical Jump Protocol (VJ) Vertical countermovement jumps will be assessed on the same force plates utilized for the MVIC. Participants will undergo 3 vertical jump trials with 1 minute rest between. Participants will be instructed to jump as high as possible with their hands on their hips. The highest value achieved in the three trials will be used to denote the participant's maximal vertical jump height. VJ will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.

Isoinertial Squat Protocol (ISP) The ISP will be conducted using the Desmotec isoinertial training device (D11 evo, Desmotec, Biella, Italy). During the ISP, participant's force and power output will be measured by the Desmotec device via two underfoot force plates. Participants will be asked to maintain a standing position with their feet at a width identical to that typically used during a traditional back squat, to cross their arms in front of them to their opposite shoulder, and to maintain that position for every ISP assessment. Participants will then be strapped into the desmotec device via the flywheel cable connected to a waist strap according to the manufacturer's instructions. Once properly fastened, cable tension will be set at 15kg using a handheld scale (ROMECH, Paisley, United Kingdom) to ensure consistent cable tautness between participants. The resulting length of each participant's cable will be recorded during V2 and standardized for all subsequent assessments. The ISP will consist of 6 sets of 10 maximal repetitions at an isoinertial resistance of .067kg/mm2. Immediately preceding each set, participants will complete two low effort "free repetitions" to prepare the participant for the rhythm of the impending isoinertial movement. Participants will be instructed to give maximal effort during the concentric (upward) phase of the movement by reaching full knee and hip extension and rocking onto the balls of their feet but to delay their braking force during the eccentric (downward) phase until the last possible moment. A rope affixed to two height adjustable stands will be positioned horizontally behind the participant to provide a reference for the end of the eccentric (downward) phase of the movement at a height that elicits a knee angle of ~90degrees when softly touched by the participant's glutes. Rope height will be established during V2 and standardized for every subsequent ISP. Participants will be instructed to repeat that squat depth for every contraction and give maximal effort throughout the entire duration of each set while being consistently verbally encouraged by the researcher.

Standardized Cool-Down Following the ISP, participants will be required to complete a dynamic cool-down by pedaling on a cycle ergometer for 3-minutes at a self-selected pace at a set resistance of 75 watts.

ELIGIBILITY:
Inclusion Criteria:

* • Male between the ages of 18-40 years old

  * Healthy, and ready for physical activity as determined by the PAR-Q+, and MHQ.
  * Participants will be required to be recreationally active (defined according to ACSM standards of at least 150 minutes exercise per week).
  * Participants will be required to have been actively resistance training for a minimum of 6 months as defined by 3 resistance training sessions per week with at least one lower body session.
  * Participants must be willing to abstain from the consumption of bananas of non-steroidal anti-inflammatory drugs (NSAIDs) for the duration of their enrollment in study.
  * Participants must be willing to abstain from dietary supplementation that are viewed by study investigators to confound the outcomes of the study (e.g., Creatine). Those currently supplementing must be willing to undergo a 28-day washout prior to beginning study procedures.
  * Participants must be consuming <300 mg·day-1 (Equivalent to 3 cups of coffee per day or 2 16oz cans of Redbull) and willing to keep their caffeine consumption consistent throughout the duration of the study.
  * Participants will be required to have access to the online MyFitnessPal application either via cellphone or computer and be willing to download and maintain the application for the duration of the study.
  * Free from previous or current lower body injuries that are viewed by the investigators to potentially limit ability of the participant to perform the assessments.
  * Willing to abstain from lower body resistance training for the 14 days preceding ET1 and ET2

Exclusion Criteria:

* • Individual does not provide consent to participate in this study.

  * Inability to perform physical exercise (determined by MHQ, and PAR Q+). That is Answering "Yes" to any question on the PAR-Q +, or having a pre-existing condition such as musculoskeletal injury, back pain, chronic pain etc. that the investigative team perceives will prevent a participant from safely completing the protocol.
  * Not currently participating in at least 150 minutes of physical activity per week.
  * Not currently resistance trained (as defined within the inclusion criteria)
  * Currently taking any performance-enhancing drug (determined from health and activity questionnaire)
  * Currently taking a nutritional supplement known to improve physical performance and not willing refrain form the consumption of the supplement for at least 28-days prior to beginning study procedures.
  * Regularly taking any type of prescription or over-the-counter medication deemed to affect performance, or having any chronic illnesses, which require medical care.
  * Have used nicotine or tobacco at any time within the last three months.
  * Report consuming bananas or NSAIDS at any time during your enrollment in the study.
  * Report daily caffeine consumption >300 mg·day-1
  * Report any lower extremity muscle soreness for visits ET1 and ET2
  * Previous or current lower body injuries viewed by the investigators to potentially limit the ability of the participant to perform the assessments.
  * Inability or unwillingness to consume the provided standardized snacks and meals in their entirety.
  * Inability or unwillingness to adhere to the diet restrictions of the study.
  * Have a food allergy to either of the two provided energy bars.
  * Inability or unwillingness to report all food and beverage consumption during the two 5-day dietary log periods.

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Venous Blood Sample Collection - Creatine Kinase | Visit 2 & visits 6-13 approx=8 weeks
  Blood samples will be obtained at V2, PRE-, IP, 24H, 48H, and 72H using a 21-gauge vacutainer or 23-gauge butterfly needle from a superficial forearm vein. Up to 2 unsuccessful attempts in one arm, and with permission, a third attempt in the opposite arm, will be made. Three failed attempts will terminate the draw. Issues with blood collection devices will not remove participants from the study. All draws will follow aseptic conditions, with skin disinfected before insertion and the puncture site bandaged afterward. A total of 8mL of blood (slightly less than 2 tsp) will be collected at each time point (V2 & V6-V13) in one 4mL BD Vacutainer™ SST. Serum tubes will be inverted, clotted at room temperature for 30 minutes, centrifuged for 10 minutes at 4000rpm, aliquoted, and frozen at -80°C within one hour. Serum will be used to determine creatine kinase (CK) concentrations, presented as U/L.
Venous Blood Sample Collection - C-Reactive protein | Visit 2 & visits 6-13 approx=8 weeks
  Blood samples at V2, PRE-, IP, 24H, 48H, and 72H will be obtained using a 21-gauge vacutainer or 23-gauge butterfly needle from a superficial forearm vein. A maximum of 2 unsuccessful attempts per arm will be allowed, with a third attempt permitted in the opposite arm if agreed upon. Three failed attempts will terminate the draw. Issues with blood collection devices will not disqualify participants from the study. All blood draws will follow aseptic conditions, with the skin disinfected before insertion and the puncture site covered with a bandage. A total of 8mL of blood (slightly less than 2 tsp) will be collected at each time point (V2 & V6-V13) in one 4mL BD Vacutainer™ SST. Serum tubes will be inverted, clotted at room temperature for 30 minutes, centrifuged for 10 minutes at 4000rpm, aliquoted, and frozen at -80°C within one hour of collection. Serum will be used to determine C-reactive protein (CRP) concentrations. and presented at U/L.
Venous Blood Sample Collection - CBC | Visit 2 & visits 6-13 approx=8 weeks
  Blood samples at V2, PRE-, IP, 24H, 48H, and 72H will be obtained using a 21-gauge vacutainer needle or 23-gauge butterfly needle from a superficial forearm vein. A maximum of two unsuccessful attempts per arm will be allowed, with a third attempt in the opposite arm if agreed upon. Three failed attempts will terminate the blood draw. Issues with blood collection devices will not disqualify participants from continuing the study. All blood draws will follow aseptic procedures, with the skin disinfected before insertion and the puncture site covered with a bandage. A total of 8mL of blood (slightly less than 2 tsp) will be collected at each time point (V2 & V6-V13) in one 4mL K2EDTA plasma tube (EDTA). EDTA samples will be analyzed same day using a Sysmex XN-450 Automated Hematology Analyzer, and used to measure hematocrit, hemoglobin, MCV, MCH, MCHC, total and differential blood cell counts, and platelets in-house at the Cellular Exercise Physiology Laboratory.
Flow Mediated Dilation (FMD) | Visit 2 & visits 6-13 approx=8 weeks
  Subjects will rest in a quiet, dimly lit laboratory in a semi-recumbent position for 15 minutes before testing. Automated sphygmomanometry will measure resting systolic blood pressure (SBP), diastolic blood pressure (DBP), and heart rate (HR) on the left arm, with mean arterial pressure (MAP) calculated. Brachial artery diameter and blood velocity will be assessed using duplex Doppler ultrasound (GE Logiq P9) with a 5-MHz transducer. A tourniquet cuff will be placed around the right forearm to induce reactive hyperemia. Baseline measurements will be recorded for 2 minutes, followed by 5 minutes of arterial occlusion at 240 mmHg, and 3 minutes post-deflation. Ultrasound settings will remain consistent, with scans performed by the same technician and saved via video capture software (Snagit). Offline analysis will use FMD Studio, with parameters calculated via custom macros in Microsoft Excel. FMD will be assessed at V2, and PRE.
Ultrasound Measurement (MT and EI) | Visit 2 & visits 6-13 approx=8 weeks
  Rectus femoris (RF), vastus medialis (VM), and vastus lateralis (VL) muscle thickness (MT) and echo intensity (EI) will be assessed on the right leg using B-mode ultrasound (GE Logiq, General Electric Medical Systems, Milwaukee, WI, USA) with a linear array probe (L4-12t, 4.2-13.0 MHz). Measurements will be performed at 12 MHz, gain of 50 dB, depth of 5 cm, and dynamic range of 72. A water-soluble gel will enhance acoustic coupling. Three images of each muscle will be captured in the sagittal plane. RF images will be taken midway between the superior patella and inguinal fold, VM images 3 inches proximal to the medial femoral epicondyle, and VL images midway between the greater trochanter and superior patella. Images will be analyzed using ImageJ software (v1.53v, NIH, Bethesda, MD) following Girts et al. (41). MT and EI will be assessed at PRE, IP, 24H, 48H, and 72H for each experimental trial.
Active Range of Motion (AROM) | Visit 2 & visits 6-13 approx=8 weeks
  AROM will be assessed following the standardized warm-up while participants are in a prone position on a padded testing table with their legs fully supported. A handheld goniometer will be used to assess AROM of the right knee. The goniometer will be anchored at the lateral epicondyle of the femur with the stationary arm in line with the greater trochanter of the femur and the movement arm aligned with the lateral malleolus of the ankle. Participants will be instructed to move the knee from maximal full extension throughout the range of motion to maximum full flexion holding each end point for two seconds. The average of two consecutive measurements will be used to determine AROM. AROM will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.
Pain Pressure Threshold | Visit 2 & visits 6-13 approx=8 weeks
  PPT will be assessed immediately following the AROM assessment while the participants sat on the end of padded table with their upper legs supported and their lower legs hanging freely. Using a handheld 15kg dolorimeter with a 1 cm rubber tip, pressure will be applied to the RF, VM, and VL at locations identical to that of the ultrasound assessments increasing at a rate of 1 kg/s until participants first report feeling pain, at which point the algometer will be removed from the skin. PPT will be assessed once at each sight before a second measure of PPT at each location is acquired. The algometer value at the onset of pain will be recorded and the average of two measures with will be used to denote PPT. PPT will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.
Perceived Recovery Scale (PRS) | Visit 2 & visits 6-13 approx=8 weeks
  PRS will be assessed as a total feeling of recovery in the lower extremities (waist down) and be performed while the participant is standing at a knee angle of 140 degrees immediately prior to MS testing. Participants will be asked to rank their level of recovery on a 100mm VAS ranging from 0 to 100, with 0 being not at all recovered and 100 being very well recovered. PRS will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.
Muscle Soreness (MS) | Visit 2 & visits 6-13 approx=8 weeks
  MS will be assessed as a total feeling of soreness in the lower extremities (waist down) and be performed while the participant is standing at a knee angle of 140 degrees immediately prior to MVIC testing. Participants will be asked to rank their level of MS of their entire lower extremities on a 100mm VAS ranging from 0 to 100, with 0 being no pain at all and 100 being the most pain imaginable. MS will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.
Maximal Voluntary Isometric Contraction (MVIC) and Rate of Force development (RFD) | Visit 2 & visits 6-13 approx=8 weeks
  MVIC assessments will be conducted using a specialized isometric squat rack with an immovable bar. Bar height, set during V2 and standardized for all subsequent assessments, will align participants to a knee angle of 140 degrees. Each MVIC session will include 3 x 5s maximal isometric contractions, where participants will drive upward against the bar by extending their knees and hips, mimicking a high bar back squat. Contractions will be initiated by a verbal prompt, with consistent encouragement provided throughout. One minute of rest will be given between contractions. The highest peak force recorded will represent the participant's MVIC, from which rate of force development (RFD) will be determined at 0-250ms from contraction onset. MVIC and RFD will be assessed at PRE, IP, 24H, 48H, and 72H during each trial.
Vertical Jump Protocol (VJ) | Visit 2 & visits 6-13 approx=8 weeks
  Vertical countermovement jumps will be assessed on the same force plates utilized for the MVIC. Participants will undergo 3 vertical jump trials with 1 minute rest between. Participants will be instructed to jump as high as possible with their hands on their hips. The highest value achieved in the three trials will be used to denote the participant's maximal vertical jump height. VJ will be assessed at PRE, IP, 24H, 48H, and 72H during each experimental trial.
Isoinertial Squat Protocol (ISP) | Visit 2 & visits 6-13 approx=8 weeks
  The ISP will be conducted using the Desmotec isoinertial training device (D11 evo, Desmotec, Biella, Italy) with force and power output measured via underfoot force plates. Participants will stand in a position mimicking a traditional back squat, arms crossed to opposite shoulders, and maintain this posture throughout. They will be strapped into the device with cable tension set to 15kg using a handheld scale (ROMECH, Paisley, UK) for consistency. Cable length will be recorded during V2 and standardized for subsequent assessments. The ISP consists of 6 sets of 10 maximal repetitions at .067kg/mm² isoinertial resistance, preceded by two low-effort "free repetitions" to establish rhythm. Participants will give maximal effort during the concentric phase, reaching full extension, and delay braking during the eccentric phase until the last moment, using a horizontal rope as a depth marker (~90° knee angle). Concentric and eccentric force and power will be averaged per set.

SECONDARY OUTCOMES:
Hydration Status | Visit 2 & visits 6-13 approx=8 weeks
  Upon arriving to the lab, participants will be given a sample cup to take to the restroom and provide a urine sample, so that hydration may be assessed. After providing a urine sample, a member of the research team will measure urine specific gravity (USG) using a refractometer to ensure participants are euhydrated (1.002-1.025). If dehydrated (>1.025), they will be asked to consume 16 oz of water and be retested after waiting 15 minutes post ingestion. If hyperhydrated (<1.002) their visits will be rescheduled. Hydration status will be checked immediately upon arrival to the laboratory for V2 and each experimental trial (V6-V13). Urine samples will be disposed of according to UCF policy.
Sleep Quality Questionnaire | Visit 2 & visits 6-13 approx=8 weeks
  Participants will be asked to fill out a brief 7 question sleep questionnaire consisting of questions pertaining to their sleep and sleep quality within the last 24 hours. Participants will complete the SQQ immediately upon arriving for each experimental trial (V6-V13)
Diet and Dietary Log | Visit 2 & visits 6-13 approx=8 weeks
  Participants will be asked to maintain two separate 5-day dietary logs using the "MyFitnessPal" application on their own cellular or computer device. Participants will be asked to begin each 5-day log 24 hours before ET1 and ET2 and to maintain the log by tracking all food and beverage consumption to the best of their ability for the 5 days until the completion of the 72H follow up visits (visits 9 & 13, respectively). Additionally, participants will be asked to keep their food and beverage consumption during the two 5-day periods as consistent as possible and to match macronutrient (fats, carbohydrates, and proteins) consumption between the two periods to the best of their ability. Participants refusing to voluntarily report food and beverage consumption will be withdrawn from the study.
Anthropometric Assessments: | Visit 2
  During V2, participants will complete anthropometric assessments of height, weight, and body composition. Height and weight will be assessed using a stadiometer and scale (Health-o-meter Professional Patient Weighing Scale, Model 500 KL, Pelstar, Alsip, IL, USA). Body composition will be assessed using bioelectrical impedance analysis (BIA; InBody 770, Biospace Co, Ltd. Seoul, Korea) or bioelectrical impedance spectroscopy analyzer (Sozo; Carlsbad, CA, USA). Participants will be asked to void their bladder, and remove shoes, socks, and all jewelry for this assessment. They will also be asked to be eight hours fasted and well-hydrated as determined by USG analysis. There are no risks or discomforts associated with the BIA analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Central Florida EPIC Lab, Orlando, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will be shared only amongst the team collecting the data as per our IRB approval.